CLINICAL TRIAL: NCT01404819
Title: Evaluation of Brain Damage Resulting From Carotid Endarterectomy With Xenon Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LOCAL/2011/JRGC; 2011-002551-33 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Carotid Endarterectomy
MeSH Terms: interventions — Anesthesia; Xenon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Patients in this arm undergo anesthesia with Xenon.
  Interventions: Drug: Anesthesia with Xenon
- Standard arm (Active Comparator): Patients in this arm undergo standard anesthesia
  Interventions: Drug: Standard anesthesia

INTERVENTIONS:
Drug: Anesthesia with Xenon — Patients undergo anesthesia with xenon (remifentanil with xenon).
  Arms: Experimental arm
Drug: Standard anesthesia — Patients undergo standard anesthesia (remifentanil with propofol)
  Arms: Standard arm

SUMMARY:
The objective of this study is to show that, in patients undergoing carotid endarterectomy, brain damage, assessed by the determination of S100B before removing the clamp, is less severe with a balanced anesthesia consisting of remifentanil combined with Xenon (experimental arm) compared with remifentanil anesthesia associated with propofol (reference arm).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patients with American Society of Anesthesiology (ASA) scores of 1 to 4
* Patient schelduled for carotid endarterectomy

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient has a contra-indication for a treatment necessary for this study
* The endarterectomy does not require a shunt
* ASA score of 5
* Patient presenting with symptomatic gastric-oesophagien reflux
* Patient has neuro-endocrine cancer
* Patient has hypersensivity to one of the following substances: propofol, remifentanil, celocurine, cisatracurium, rocuronium, senon, paracetamol, tramadol
* Patient suffering from obstructive respiratory insufficiency (chronic obstructive pulmonary disease, asthma)
* Patient with coronary disease with severely altered cardiac function
* High intracranial pressure
* Patient requiring high concentrations of oxygen (SpO2 < 92% normal air)
* Patient with neuro-sensorial deficit that, in the absence of a prothesis, prevents reading, writing, or responding to simple orders
* Patient suffering from myopathy or recent rhabdomyolysis
* Patient with psychiatric pathology or chronic alcohol consumption or consumption of another substance that interferes with understanding
* Lack of contraception for women of child-bearing age
* History of or suspected malignant hyperthermia
* Patients with liver damage, jaundice, unexplained fever or eosinophilia after administration of a halogenated anesthetic
* Patient has undergone a recent multiple trauma (<1 month)
* Patient who received general anesthesia within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Presence/absence of S100B > 0.2 ng/ml during surgery | During surgery (expected mean time of around 120 minutes)
  Presence/absence of S100 calcium binding protein B concentration after induction and before the removal of the radial arterial catheter clamp placed before induction

SECONDARY OUTCOMES:
S100B change relative to baseline | end of surgery (expected mean of 120 minutes)
  The change in S100 calcium binding protein B concentration before and after surgery (ng/ml)
NSE change from baseline | end of surgery (expected mean of 2 hours), just before clamp removal
  The change in Neuron Specific Enolase (NSE) between a preoperative measurement and a second measurement near the end of surgery and just before clamp removal
NSE change from baseline | end of surgery (expected mean of 2 hours)
  The change in Neuron Specific Enolase (NSE) between a preoperative measurement and a second measurement just after surgery
Change in troponine from baseline | end of surgery (expected mean of 2 hours)
  Change in tropinine between preoperative and postoperative measurements
Change in creatinemia from baseline | end of surgery (expected mean of 2 hours)
  Change in creatinemia between preoperative and postoperative measurements
Change in creatine clearance from baseline | end of surgery (expected mean of 2 hours)
  Change in creatine clearance (MDRD equation) between preoperative and postoperative measurements
Change NIHSS score from baseline | end of surgery (expected mean of 2 hours)
  Change in the National Institute of Health Stroke Score (NIHSS) between preoperative and postoperative measurements
Number of transfusions | During surgery (estimated mean of 120 minutes)
  Number of transfused red blood cell packs
Direct costs | 2 days
  Direct costs (€) incurred
Indirect costs | 2 days
  The indirect costs (€) incurred

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ripart, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France